CLINICAL TRIAL: NCT03507595
Title: Evaluation of the Metastasis and Recurrence of Prostate Cancer With 18F-PSMA PET/CT
Brief Title: Evaluation of the Metastasis and Recurrence of Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-17-020
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2017-12

CONDITIONS: Prostate Cancer (Diagnosis); Prostate Cancer Metastatic; Prostate Cancer Recurrent; Prostate Cancer Stage
Keywords: prostate specific membrane antigen(PMSA); prostate cancer; PET/CT
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with initial diagnosis of PCa: 1. T2 stage: PSA>20ng/ml, Gleason Score >= 8;
  2. T3 or T4 stage;
  3. The imaging examination was negative or localized metastasis of the pelvic lymph node, but there was no distant metastasis of lymph nodes or bone and internal organs other than the pelvic cavity.
- Patients with biochemical recurrent PCa: 1. After the RRP surgery,the serum PSA was over 0.2 ng/ml in two consecutive sera;
  2. After the radiotherapy: the lowest PSA is up to 2 ng/ml.
- Patients with CRPC: 1. The serum testosterone is in the castration level (< 50 ng/dL or < 1.7 nmol/L);
  2. The PSA is elevated 3 times in a row, the base value is increased by more than 50%, and the PSA > 2ng/mL(the interval is one week);
  3. The continuation of the anti-androgen drugs, flunamine was stopped for at least 4 weeks, and biglumide was suspended for at least 6 weeks;
  4. Despite the continued standard androgen deprivation therapy, the PSA is still progressing.

SUMMARY:
This study aims to use the new molecular probe 18F-PSMA for the diagnosis,staging ,recurrence monitoring and evaluation of the prostate cancer.By compared with the conventional imaging methods (whole body bone scintigraphy and MRI) and molecular imaging methods (11C-choline PET/CT),we hope to find the advantages of 18F-PSMA PET/CT in the diagnosis and metastases of prostate cancer, and lay the foundation for the further clinical transformation.

DETAILED DESCRIPTION:
This study aims to use the new molecular probe 18F-PSMA for the diagnosis,staging ,recurrence monitoring and evaluation of the prostate cancer.By compared with the conventional imaging methods (whole body bone scintigraphy and MRI) and molecular imaging methods (11C-choline PET/CT),we hope to find the advantages of 18F-PSMA PET/CT in the diagnosis and metastases of prostate cancer, and lay the foundation for the further clinical transformation.And make some comparison with those 3 methods.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with initial diagnosis of prostate cancer; 1）T2 stage: PSA>20ng/ml, Gleason Score >= 8; 2）T3 or T4 stage; 3）The imaging examination was negative or localized metastasis of the pelvic lymph node, but there was no distant metastasis of lymph nodes or bone and internal organs other than the pelvic cavity.
2. Patients with biochemical recurrent prostate cancer; 1）After the RRP surgery, the serum PSA was over 0.2 ng/ml in two consecutive sera; 2）After the radiotherapy: the lowest PSA is up to 2 ng/ml.
3. Patients with CRPC. 1）The serum testosterone is in the castration level (< 50 ng/dL or < 1.7 nmol/L); 2）The PSA is elevated 3 times in a row, the base value is increased by more than 50%, and the PSA > 2ng/mL(the interval is one week); 3）The continuation of the anti-androgen drugs, flunamine was stopped for at least 4 weeks, and biglumide was suspended for at least 6 weeks; 4）Despite the continued standard androgen deprivation therapy, the PSA is still progressing.

Exclusion Criteria:

1. Patients who are unwilling to participate in the study or unwilling to sign the informed consent forms;
2. Patients who are critically ill, suffering from mental illness and cannot cooperate with the examination;
3. There are electronic implants, such as pacemakers and insulin pumps in the body, and magnetic metal foreign objects in the spot.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Aged male
Study Population: * Patients with initial diagnosis of prostate cancer;
  * Patients with biochemical recurrent prostate cancer;
  * Patients with CRPC.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
18F-PSMA PET/CT imaging | 4 hours
  The outcome of 18F-PSMA PET/CT imaging.

SECONDARY OUTCOMES:
Bone scan imaging | 6 hours
  The outcome of bone scan imaging.
MRI imaging | 4 hours
  The outcome of MRI imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Hongliang Fu, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT03507595/ICF_000.pdf